CLINICAL TRIAL: NCT04304612
Title: A Cost Effective and Time Saving Blood Test to Detect Six Human Bloodborne Infectious Diseases (SAFE-Blood)
Brief Title: A Cost Effective and Time Saving Blood Test to Detect Six Human Bloodborne Infectious Diseases
Acronym: SAFE-Blood
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0141
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: HIV; Viral Hepatitis
Keywords: Serological assays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Samples without DNA : Three sample collections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The consortium will develop a new in vitro diagnostic (IVD) test to screen donated blood for bloodborne infectious pathogens, saving blood banks time and costs required for analysis of mandatory pathogens. The IVD test is a multiplex immunoassay that simultaneously screens for six bloodborne infectious diseases per blood sample. In this project, a mix of diagnostic protein markers will be developed and validated to lowdown an IVD test ready for commercial scale-up and CE-IVD certification.

ELIGIBILITY:
Inclusion criteria:

- Samples having been tested positive or negative for the serological markers explored in the study

Exclusion criteria:

- to refuse to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collection of human biological samples integrated into the laboratory's declared collections. These samples come from major subjects taken as part of a diagnostic or monitoring procedure for infection with viral hepatitis or HIV
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Analytical performances | day 1
  Analytical performances

SECONDARY OUTCOMES:
Number of Field evaluation | day 1
  Field evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Edouard TUAILLON, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC